CLINICAL TRIAL: NCT07269691
Title: RaSOLVE: An Open-Label, Controlled, Randomized, Multicenter Phase III Clinical Trial Assessing the Impact of Preoperative 125I Radioactive Seed Localization on Pathological Complete Response Rate (tpCR: ypT0/is ypN0) and Long-Term Prognosis (iDFS/OS) in Women With Early or Locally Advanced Newly Diagnosed Untreated Breast Cancer Following Neoadjuvant Therapy
Brief Title: RaSOLVE: 125I Radioactive Seed Marking Effects on Pathological Complete Response Rate and Prognosis Post-Neoadjuvant Therapy in Early/Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pengfei Qiu (Other)
Responsible Party: Sponsor-Investigator, Pengfei Qiu, Chief Physician, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-477-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Breast Cancer
Keywords: Iodine-125 seed Radioactive seed marking Breast cancer Neoadjuvant therapy Pathological complete response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to the iodine-125 seed marking group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iodine-125 Seed Marking (Experimental): Participants in this arm will undergo ultrasound-guided implantation of Iodine-125 radioactive seeds (0.1-0.3 mCi) into the primary breast tumor and biopsy-confirmed metastatic axillary lymph nodes before starting neoadjuvant therapy. Seed position will be monitored every two cycles using ultrasound and confirmed preoperatively by mammography and MRI. After implantation, all participants will receive standard neoadjuvant therapy followed by surgery and pathological assessment according to study protocol.
  Interventions: Device: Iodine-125 Radioactive Seed Marking; Drug: Standard Neoadjuvant Therapy
- No Seed Marking (Active Comparator): Participants in this arm will receive standard neoadjuvant therapy without implantation of iodine-125 seeds. After neoadjuvant therapy is completed, participants will undergo surgery and pathological evaluation according to standard clinical practice.
  Interventions: Drug: Standard Neoadjuvant Therapy

INTERVENTIONS:
Device: Iodine-125 Radioactive Seed Marking — Ultrasound-guided implantation of iodine-125 radioactive seeds (0.1-0.3 mCi) into the primary breast tumor and biopsy-confirmed positive axillary lymph nodes prior to the first cycle of neoadjuvant therapy. Seed position will be verified during treatment using ultrasound, mammography, and MRI.
  Arm(s) Applied to：
  Arms: Iodine-125 Seed Marking
Drug: Standard Neoadjuvant Therapy — Systemic neoadjuvant therapy based on breast cancer subtype and clinical guidelines, which may include chemotherapy, targeted therapy, immunotherapy, or endocrine therapy as assessed by investigators. All participants in both arms will receive neoadjuvant therapy followed by surgery.

SUMMARY:
This study is an open-label, controlled, multicenter phase III clinical trial designed to evaluate whether the use of iodine-125 radioactive seed markers can improve treatment response for patients with early or locally advanced breast cancer undergoing neoadjuvant therapy.

Neoadjuvant therapy is widely used for breast cancer to shrink tumors, increase the chances of breast-conserving surgery, and help determine the most effective postoperative treatments. Achieving a pathological complete response (pCR) after neoadjuvant therapy is strongly associated with better long-term outcomes.

In this study, qualified participants will be randomly assigned in a 1:1 ratio to either the experimental group or the control group.

Experimental group: Patients will receive placement of iodine-125 seed markers in the primary breast tumor and biopsy-proven positive axillary lymph nodes before starting neoadjuvant therapy.

Control group: Patients will undergo standard neoadjuvant therapy without seed placement.

All participants will then complete neoadjuvant therapy followed by surgery. Pathological evaluation will determine whether the cancer has completely disappeared. Long-term outcomes, including invasive disease-free survival, will be followed for at least five years.

The goal of this study is to determine whether radioactive seed marking can increase the rate of pathological complete response and improve prognosis in patients receiving neoadjuvant therapy for breast cancer. The study will also explore whether iodine-125 seeds may activate immune responses that contribute to treatment effectiveness.

DETAILED DESCRIPTION:
This multicenter, open-label, controlled phase III clinical trial aims to investigate the clinical value of iodine-125 radioactive seed markers in patients with early or locally advanced breast cancer undergoing neoadjuvant therapy. Current guidelines support pre-treatment marking of primary tumors and lymph nodes to improve surgical accuracy and reduce false-negative rates in sentinel lymph node biopsy after neoadjuvant therapy. However, the optimal marking method remains unclear. Iodine-125 seeds offer potential advantages, including high localization accuracy, improved identification of metastatic lymph nodes, and favorable cost-effectiveness compared with other wireless or metallic markers.

Eligible patients will be randomized 1:1 into either the experimental or control group.

Experimental group: Under ultrasound guidance, iodine-125 seeds (0.1-0.3 mCi) will be implanted into the primary breast tumor and biopsy-proven positive axillary lymph nodes before the first cycle of neoadjuvant therapy. Seed positions will be monitored throughout therapy by ultrasound, mammography, and MRI to confirm they have not migrated (defined as ≤5 mm deviation from baseline).

Control group: Patients will receive neoadjuvant therapy without seed implantation.

All participants will receive standard neoadjuvant systemic therapy according to disease subtype and investigator assessment. Following therapy, participants will undergo surgery, and pathological responses will be evaluated by predefined criteria. Patients will be followed for at least five years to assess invasive disease-free survival and other outcomes.

Objectives and Endpoints

The primary objective is to compare the pathological complete response (pCR) rate between the seed-marked arm and the control arm. pCR is defined as ypT0/is and ypN0, meaning no residual invasive carcinoma in the breast or regional lymph nodes.

Secondary objectives include breast pCR (bpCR), axillary pCR (apCR), and invasive disease-free survival (iDFS). An exploratory endpoint will evaluate whether iodine-125 seeds may stimulate immune activation by monitoring peripheral blood CD4+/CD8+ T-cell ratios during treatment.

Study Rationale

Neoadjuvant therapy plays a critical role in downstaging tumors and improving surgical options. Achieving pCR is associated with significantly improved long-term survival outcomes, particularly for HER2-positive and triple-negative breast cancer. Our preliminary work suggests that patients receiving iodine-125 seed implantation prior to neoadjuvant therapy show improved pCR rates across molecular subtypes compared with patients without seed placement. Therefore, this trial aims to confirm the effectiveness and safety of radioactive seed marking in a rigorously controlled phase III study and to explore its biological mechanisms.

Safety Monitoring

Adverse events and serious adverse events will be recorded from the time informed consent is obtained until postoperative follow-up. All safety assessments, including laboratory tests, imaging, and clinical examinations, will be performed according to protocol-defined schedules. The relationship between adverse events and seed implantation will be evaluated by investigators following prespecified criteria.

This trial is expected to provide high-quality evidence regarding the clinical utility of iodine-125 seeds in improving response assessment, enhancing pCR rates, and potentially affecting long-term prognosis in breast cancer patients receiving neoadjuvant therapy. It may also contribute novel insights into radiotherapy-related immunomodulatory mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 70 years.
* ECOG performance status 0-1.
* Pathologically confirmed, previously untreated, unilateral primary invasive breast cancer.
* Clinical stage cT1cN1-2M0 or cT2-3N0-2M0 (AJCC 8th edition).
* Adequate organ function within 7 days prior to randomization:

  * Hemoglobin ≥ 90 g/L
  * ANC ≥ 1.5×10⁹/L; Lymphocyte count ≥ 0.5×10⁹/L
  * Platelet count ≥ 100×10⁹/L
  * WBC 3.0-15×10⁹/L
  * ALT, AST ≤ 2.5×ULN; ALP ≤ 2.5×ULN; TBIL ≤ 1.5×ULN
  * Serum creatinine ≤ 1.5×ULN and creatinine clearance ≥ 60 mL/min
  * PT, APTT ≤ 1.5×ULN
  * Urine protein < 2+ or 24-hour urine protein ≤ 1 g
  * LVEF ≥ 55%
  * QTcF < 470 ms
* Negative serum pregnancy test within 3 days prior to first treatment for women of childbearing potential and agreement to use effective contraception.
* Willing and able to sign informed consent.

Exclusion Criteria:

* Bilateral breast cancer or history of DCIS, LCIS, invasive breast cancer, or metastatic breast cancer.
* Any malignancy diagnosed within the past 5 years except cured cervical carcinoma in situ or non-melanoma skin cancer.
* Prior systemic chemotherapy, targeted therapy, immunotherapy, or radiotherapy within 1 year.
* Prior exposure to anthracyclines, taxanes, or platinum agents.
* Primary or secondary immunodeficiency; uncontrolled autoimmune disease (except controlled hypothyroidism or type 1 diabetes).
* Interstitial lung disease or severe chronic lung disease.
* Clinically significant cardiovascular disease, including:

  * NYHA class ≥ III
  * Myocardial infarction or stroke within 3 months
  * Uncontrolled hypertension
  * Clinically significant arrhythmia or heart failure
* Arterial/venous thrombosis within 3 months.
* Vaccination with live attenuated vaccine within 28 days.
* Active HBV, HCV, or HIV infection.
* Major surgery within 28 days (except diagnostic procedures).
* Severe infection within 4 weeks or systemic antibiotic-treated infection within 2 weeks.
* History of bone marrow or organ transplantation.
* Coagulation abnormalities (INR > 1.5 or APTT > 1.5×ULN).
* Peripheral neuropathy ≥ Grade 2.
* Treatment with systemic immunostimulatory agents within 4 weeks or immunosuppressive agents within 2 weeks.
* Known allergy to study agents.
* Participation in another clinical trial within 4 weeks.
* Pregnancy, breastfeeding, or planning pregnancy.
* Substance abuse or psychiatric conditions that may affect compliance.
* Any condition that, in the investigator's judgment, makes the patient unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | At the time of surgery, approximately 6-8 months after enrollment
  Pathologic complete response (pCR) is defined as no residual invasive carcinoma in both the resected breast tissue and ipsilateral regional lymph nodes following completion of neoadjuvant therapy and surgery (ypT0/is, ypN0). Residual ductal carcinoma in situ (DCIS) may be present. This definition is fully consistent with the study protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive clinical information and is subject to institutional and regulatory restrictions in China. Data sharing is not planned due to privacy protection requirements and limitations in the current data management framework.